CLINICAL TRIAL: NCT03154333
Title: An International, Multicenter, Randomized, Double-Blind, Parallel-Group Phase 2 Study Evaluating the Safety and Efficacy of Diacerein 1% Ointment Topical Formulation in Subjects With Epidermolysis Bullosa Simplex
Brief Title: Safety and Efficacy of Diacerein 1% Ointment for Subjects With Epidermolysis Bullosa Simplex (EBS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Castle Creek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCP-020-301
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Epidermolysis Bullosa Simplex
Keywords: Epidermolysis; bullosa; simplex; EBS
MeSH Terms: conditions — Epidermolysis Bullosa Simplex | interventions — diacerein; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- diacerein 1% ointment (Experimental): diacerein 1% ointment will be used for 8 weeks
  Interventions: Drug: diacerein 1% ointment
- vehicle ointment (Placebo Comparator): vehicle ointment will be used for 8 weeks
  Interventions: Drug: A placebo ointment

INTERVENTIONS:
Drug: diacerein 1% ointment — diacerein 1% ointment administered topically
  Other Names: CCP-020
  Arms: diacerein 1% ointment
Drug: A placebo ointment — vehicle ointment administered topically
  Arms: vehicle ointment

SUMMARY:
Epidermolysis bullosa simplex (EBS) is a rare genetic skin disease characterized by fragility of the skin and mucous membranes resulting in painful blisters and erosions after minor trauma. The purpose of this study is to compare the efficacy of diacerein 1% ointment to vehicle ointment when applied once-daily for 8 weeks in subjects with EBS.

DETAILED DESCRIPTION:
The study is an international, multicenter, randomized, double-blind, vehicle-controlled, parallel group study to evaluate the safety and efficacy of diacerein 1% ointment for the treatment of subjects with EBS. Participants were assigned to study groups receiving either diacerein 1% ointment or vehicle ointment for 8 weeks, followed by an 8 week follow-up period. Approximately 80 subjects were to be randomized to one of the 2 treatment groups.

The primary objective of this study is to compare the efficacy of diacerein 1% ointment to vehicle ointment based on reduction in body surface area (BSA) of EBS lesions being treated when applied once-daily for 8 weeks in subjects with EBS. The secondary objectives are to compare the effects of diacerein 1% ointment to vehicle ointment in subjects with EBS in changes in Investigator Global Assessment (IGA) scores, pain, pruritus, mobility, and safety and tolerability.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is at least 4 years of age at Screening
* Subject has a documented genetic mutation consistent with EBS. Gene mutations acceptable for inclusion are as follows: KRT5, KRT14, PLEC1, TGM5, PKP1, DSP, FERMT1, EXPH5, DST, KLHL24.
* Subject has an Assessment Area of EBS lesions to be treated, that is ≥2% body surface area (BSA) and the EBS lesions are in one or both of the following body areas:

  * Localized: plantar and/or palmar areas
  * Generalized: arms, legs, torso, hands and feet
* Subject's EBS lesions in the Assessment Area have an Investigator's Global Assessment (IGA) score of ≥3
* Subject/caregiver agrees to not use any topical therapies other than the study medication that might influence the status of the EBS lesions during the duration of the study
* Subject is non-pregnant as confirmed by a negative urine pregnancy screen, non-lactating and is not planning for pregnancy during the study period
* If the subject is a woman of childbearing potential, agrees to use an approved effective method of birth control
* Subject is in good general health and free of any known disease state or physical condition which might impair evaluation of the EBS lesions or which exposes the subject to an unacceptable risk by study participation

Key Exclusion Criteria:

* Subject has EBS lesions to be treated that are infected
* Subject has used any diacerein containing product within 6 months prior to Screening
* Subject has used systemic immunotherapy or cytotoxic chemotherapy within 60 days prior to Screening
* Subject has used systemic steroidal therapy or has used topical steroidal therapy on the EBS lesions to be treated within 30 days prior to Baseline
* Subject has evidence of a systemic infection or has used systemic antibiotics within 7 days prior to Screening
* Subject is currently using systemic analgesics and/or anti-histamine therapy, for treatment of EBS lesions unless on a stable regimen (i.e., the same dosing regimen) for at least 4 weeks prior to Screening
* Subject has used any systemic diuretics or cardiac glycosides or any systemic product that might put the subject at undue risk
* Subject has used any topical product containing allantoin on the EBS lesions to be treated within 30 days prior to Screening
* Subject has a current malignancy, or a history of treatment for a malignancy within 2 years prior to Screening
* Subject currently has diabetes mellitus (HbA1c ≥6.5%) or controlled diabetes (HbA1c < 6.5%)
* Subject has a history of cardiac, hepatic (ALT and or AST >2x ULN, Total bilirubin >1.5x ULN at Screening), or renal disease (eGFR<30 ml/min/1.73 m^2)
* Subject has a non-EBS skin disease or condition (e.g., sunburn) that might put the subject at undue risk by study participation or interferes with the study medication application or the study assessments

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Director — Castle Creek Pharmaceuticals
Locations (22):
- United States (12):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri Healthcare, Columbia, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Children's Hospital of San Antonio ; Texas Dermatology and Laser Specialists, San Antonio, Texas
- Premier Specialists Pty Ltd; The Church, Kogarah, New South Wales, Australia
- EB House Austria, Salzburg, Austria
- France (3):
  - Hopital Saint Louis, Paris, Cedex
  - Hopital Necker-Enfants Malades, Paris, Cedex
  - CHU de NICE - Hopital de l'Archet II - Service de Dermatologie, Nice
- University Medical Center Freiburg, Freiburg im Breisgau, Germany
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- University Medical Center Groningen, Groningen, Netherlands
- United Kingdom (2):
  - Great Ormond Street Hospital, London, England
  - St. Thomas' Hospital - St Johns Institute of Dermatology, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Ointment: vehicle ointment will be used for 8 weeks
  vehicle ointment administered topically
Period: Overall Study
Arm/Group | Diacerein 1% Ointment | Vehicle Ointment
Started | 28 | 26
Completed | 21 | 21
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Population: All efficacy endpoints were based on the Assessment Area, defined in the protocol, unless otherwise stated. The Intent to Treat (ITT) Population was used for these analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diacerein 1% Ointment | Vehicle Ointment | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Customized [Count of Participants; unit: Participants]
  Age <8 years old | 13 | 12 | 25
  Age greater than or equal to 8 years old | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Baseline BSA(Body Surface Area) of EBS(Epidermolysis Bullosa Simplex) Lesions within Assessment Area [Mean (Standard Deviation); unit: Percent of BSA] | 5.76 (4.674) | 7.13 (7.606) | 6.42 (6.237)
Baseline IGA Score of 3 or 4 [Count of Participants; unit: Participants] — The investigator's global assessment (IGA) is a five-point scale that is used for overall clinical assessment of severity of disease and classifies EBS-involved skin with a score ranging from 0-4, with higher numbers indicating more severe disease.
  Participants
    IGA Score: 3 | 26 | 24 | 50
    IGA Score: 4 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieved ≥ 60% Reduction in Body Surface Area (BSA) of EBS Lesions Within Assessment Area
Description: Analysis of the proportion of subjects who achieved a ≥60% reduction in Body Surface Area (BSA) of EBS lesions within Assessment Area from Baseline to Week 8
Time Frame: Baseline to Week 8
Population: All efficacy analyses were conducted using the Intent to Treat (ITT) Population that consisted of all randomized subjects who were dispensed study drug. Subjects were included in the treatment group to which they were assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Diacerein 1% Ointment | Vehicle Ointment
Number analyzed (Participants) | 28 | 26
Participants | 16 | 14
Statistical Analysis 1: Comparison: Diacerein 1% Ointment vs Vehicle Ointment; Test type: Other; p = 0.9666, Cochran-Mantel-Haenszel; Log transformation normalized the Risk Ratio (RR) estimates; the Standard Error (SE) of the estimate was obtained from confidence limits for the RR; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.63 to 1.62]

2. Secondary Outcome: The Proportion of Subjects Who Achieved Success on the Investigator's Global Assessment (IGA)
Description: The investigator's global assessment (IGA) is a five-point scale that is used for overall clinical assessment of severity of disease and classifies EBS-involved skin with a score ranging from 0-4. Success on the IGA was defined as ≥2-point reduction from Baseline to Visit 6 (Week 8).
  IGA Scoring:
  0 = Clear; 1 = Near Clear; 2 = Mild; 3 = Moderate; 4 = Severe
  Minimum score = 0 Maximum score = 4; higher score = worse outcome
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Diacerein 1% Ointment: diacerein 1% ointment will be used for 8 weeks
  diacerein 1% ointment: diacerein 1% ointment administered
Arm/Group | Diacerein 1% Ointment | Vehicle Ointment
Number analyzed (Participants) | 28 | 26
Participants | 12 | 7
Statistical Analysis 1: Comparison: Diacerein 1% Ointment vs Vehicle Ointment; Test type: Other; p = 0.2861, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.53, 95% CI 2-sided [0.41 to 3.28]

ADVERSE EVENTS:
Time Frame: Baseline to Week 16
Arm/Group | Diacerein 1% Ointment | Vehicle Ointment
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 2/26
Other Adverse Events (participants affected / at risk) | 16/28 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diacerein 1% Ointment (N=28) | Vehicle Ointment (N=26)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniere's Disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diacerein 1% Ointment (N=28) | Vehicle Ointment (N=26)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Skin Infection (Infections and infestations) | 3 (4) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Application Site Pruritus (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT03154333/SAP_000.pdf
  • Study Protocol (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03154333/Prot_001.pdf